CLINICAL TRIAL: NCT01022008
Title: Respiratory Improvement of Faciocraniosynostosis by Craniofacial Osteodistraction
Brief Title: Assessment Study of Faciocraniosynostosis by Craniofacial Osteodistraction
Acronym: CRANIORESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: K071202
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Faciocraniosynostoses
Keywords: Exorbitism; Upper respiratory airways; Osteodistraction; Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Osteodistraction techniques (Experimental): Osteodistraction techniques
  Interventions: Device: Osteodistraction techniques

INTERVENTIONS:
Device: Osteodistraction techniques — Treatment based on craniofacial osteotomies and osteodistraction techniques.

SUMMARY:
Context. Faciocraniosynostoses present with an insufficient growth of the craniofacial skeleton due to premature fusion of skull and facial sutures. There are prenatal conditions with functional (risk of raised intracranial pressure) and morphological consequences (exorbitism, and impairment of upper respiratory airways), the severity of which justifies an early surgical treatment based on craniofacial osteotomies and osteodistraction techniques.

Distraction techniques were started in our unit eleven years ago, and never ceased to be modified: Recent improvements allowed better correction of exorbitism and therefore reduction of visual risks. But the improvements of the respiratory function remain insufficient. The initial evaluations of the respiratory functions were based on blood oxygenation monitoring, and showed real improvement. But we have routinely screened our patients with complete polysomnography examinations for the past year, and this has always revealed the existence of severe sleep apnea syndromes that we fail to correct completely, although there were slightly improved.

The aim of this PHRC protocol is :

* the qualitative and quantitative improvement of the respiratory status with a reinforced task force group including the specialists in genuine multidisciplinary approach.
* A modification of the surgical technique including modifications of the existing distraction devices, an increased number of implanted devices, and maybe a change in the surgical strategy.

DETAILED DESCRIPTION:
Study design. This is a monocentric study, the patient being its own control. Due to the extremely low incidence of these conditions, it is foreseen to include twelve patients per year, during two years, which represent 24 patients in total with a minimum follow-up of one year.

Evaluation criteria. The main evaluation criteria are the polysomnography variables (sleep apnea index, characterization of obstructive versus central respiratory events, the oxygenation pattern through the night), which will be performed before and after surgery (6 and 12 months post-op). The secondary criteria are the exorbitism correction analysed with the globe protrusion index and the rate of infections. A multidisciplinary task force group has already been structured in Necker Hospital.

Expected results. We expect to analyze and correct all the sleep apnea syndromes. Many modifications could be made on the distractors, including removal of the activation rods, bioresorbable parts, as well as the modification of the surgical techniques.

ELIGIBILITY:
Inclusion Criteria:

* age under 18 years
* faciocraniosynostosis
* surgery indication to craniofacial osteotomies
* informed consent
* social security

Exclusion Criteria:

* no possibilities of follow-up during one year post-surgery
* history of radiotherapy
* acquired or hereditary immunodeficiency syndromes
* mental retardation
* bone conditions could not support distractors

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2009-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Improvement of respiratory function | 6 months and 1 year

SECONDARY OUTCOMES:
Otorhinolaryngology events | 6 months and one year
Post-surgery infections | post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eric Arnaud, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Necker, Paris, France

REFERENCES:
- [Result] Khonsari RH, Haber S, Paternoster G, Fauroux B, Morisseau-Durand MP, Cormier-Daire V, Legeai-Mallet L, James S, Hennocq Q, Arnaud E. The influence of fronto-facial monobloc advancement on obstructive sleep apnea: An assessment of 109 syndromic craniosynostoses cases. J Craniomaxillofac Surg. 2020 Jun;48(6):536-547. doi: 10.1016/j.jcms.2020.04.001. Epub 2020 Apr 13. PMID 32354613